CLINICAL TRIAL: NCT02373202
Title: A Randomized, Double-blind, Multicenter Study Evaluating the Safety and Efficacy of Sarilumab Added to Non-MTX DMARDs or as Monotherapy in Japanese Patients With Active Rheumatoid Arthritis
Brief Title: A Study Assessing the Safety and Efficacy of Sarilumab Added to Non-MTX DMARDs or as Monotherapy in Japanese Patients With Active Rheumatoid Arthritis (SARIL-RA-HARUKA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTS13618; U1111-1160-6525 (Other: UTN)
Record Dates: First submitted 2015-02-12; First posted 2015-02-26 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; Sulfasalazine; Leflunomide; bucillamine; Tacrolimus; mizoribine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: Yes

ARMS (4):
- Sarilumab 150 mg q2w + DMARDs (Experimental): Participants received sarilumab 150 mg, subcutaneous (SC) injection, once every two weeks (q2w) along with non-MTX DMARDs (sulfasalazine, leflunomide, bucillamine, tacrolimus, and/or mizoribine) for up to 52 weeks.
  Interventions: Drug: Sarilumab; Drug: Sulfasalazine; Drug: Leflunomide; Drug: Bucillamine; Drug: Tacrolimus; Drug: Mizoribine
- Sarilumab 200 mg q2w + DMARDs (Experimental): Participants received sarilumab 200 mg, SC injection, q2w along with non-MTX DMARDs (sulfasalazine, leflunomide, bucillamine, tacrolimus, and/or mizoribine) for up to 52 weeks.
  Interventions: Drug: Sarilumab; Drug: Sulfasalazine; Drug: Leflunomide; Drug: Bucillamine; Drug: Tacrolimus; Drug: Mizoribine
- Sarilumab 150 mg q2w (Experimental): Participants received sarilumab 150 mg, SC injection, q2w for up to 52 weeks.
  Interventions: Drug: Sarilumab
- Sarilumab 200 mg q2w (Experimental): Participants received sarilumab 200 mg, SC injection, q2w for up to 52 weeks.
  Interventions: Drug: Sarilumab

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form:solution
  Other Names: SAR153191 (REGN88)
Drug: Sulfasalazine — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Sarilumab 150 mg q2w + DMARDs; Sarilumab 200 mg q2w + DMARDs
Drug: Leflunomide — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Sarilumab 150 mg q2w + DMARDs; Sarilumab 200 mg q2w + DMARDs
Drug: Bucillamine — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Sarilumab 150 mg q2w + DMARDs; Sarilumab 200 mg q2w + DMARDs
Drug: Tacrolimus — Pharmaceutical form: Capsule Route of administration: Oral
  Arms: Sarilumab 150 mg q2w + DMARDs; Sarilumab 200 mg q2w + DMARDs
Drug: Mizoribine — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Sarilumab 150 mg q2w + DMARDs; Sarilumab 200 mg q2w + DMARDs

SUMMARY:
Primary Objective:

To document the long-term safety of sarilumab added to non-methotrexate (non-MTX) disease-modifying antirheumatic drugs (DMARDs) or as monotherapy.

Secondary Objective:

To document the long term efficacy of sarilumab added to non-MTX DMARDs or as monotherapy.

DETAILED DESCRIPTION:
Total study duration was up to 62 weeks: Up to 4-week screening period, 52-week treatment period, and 6-week post-treatment follow-up period.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of rheumatoid arthritis (RA), according to the American College of Rheumatology/The European League Against Rheumatism (ACR/EULAR) 2010 Rheumatoid Arthritis Classification Criteria with >=3 months disease duration.

Moderately to severely active RA defined as:

* At least 4 of 68 tender joints and 4 of 66 swollen joints at screening visit.
* High sensitivity C-Reactive Protein (hs-CRP) >=4 mg/L or Erythrocyte Sedimentation Rate (ESR) >=28 mm/hr at screening visit.

For the combination stratum:

Participants who had continuous treatment with non-biologic DMARDs other than MTX for at least 12 weeks prior to the randomization and on a stable dose for a minimum of 6 weeks prior to screening.

For the monotherapy stratum:

Participants who per investigator judgment were any of inappropriate, intolerant or inadequate to MTX treatment.

Exclusion criteria:

Participants <20 years of age. Prior treatment with tumor necrosis factor (TNF) antagonists or any other RA-directed biologic agents without the appropriate off-drug period prior to screening.

Prior treatment with anti-interleukin-6 (anti-IL-6) or anti-interleukin-6 receptor (IL-6R) antagonist therapies, including but not limited to tocilizumab or sarilumab.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (40):
- Japan (40):
  - Investigational Site Number 392010, Asahi-Shi
  - Investigational Site Number 392001, Asahikawa-Shi
  - Investigational Site Number 392070, Beppu-Shi
  - Investigational Site Number 392036, Chiba
  - Investigational Site Number 392083, Chūōku
  - Investigational Site Number 392004, Fukui-shi
  - Investigational Site Number 392039, Fukuoka
  - Investigational Site Number 392030, Ichinomiya-Shi
  - Investigational Site Number 392002, Iizuka-Shi
  - Investigational Site Number 392019, Kagoshima
  - Investigational Site Number 392066, Kamakura-Shi
  - Investigational Site Number 392050, Kato-Shi
  - Investigational Site Number 392037, Kawachi-Nagano-Shi
  - Investigational Site Number 392099, Kawasaki-Shi
  - Investigational Site Number 392013, Kitakyushu-Shi
  - Investigational Site Number 392097, Kochi
  - Investigational Site Number 392065, Kushiro
  - Investigational Site Number 392026, Matsuyama
  - Investigational Site Number 392034, Miyagi-Gun
  - Investigational Site Number 392076, Nagoya
  - Investigational Site Number 392080, Nagoya
  - Investigational Site Number 392046, Narashino-Shi
  - Investigational Site Number 392062, Okayama
  - Investigational Site Number 392027, Osaki-Shi
  - Investigational Site Number 392059, Ōita
  - Investigational Site Number 392049, Sagamihara-Shi
  - Investigational Site Number 392014, Sapporo
  - Investigational Site Number 392041, Sapporo
  - Investigational Site Number 392073, Sapporo
  - Investigational Site Number 392006, Sasebo-Shi
  - Investigational Site Number 392021, Sendai
  - Investigational Site Number 392022, Sendai
  - Investigational Site Number 392033, Sendai
  - Investigational Site Number 392071, Sendai
  - Investigational Site Number 392029, Shizuoka
  - Investigational Site Number 392023, Takaoka-Shi
  - Investigational Site Number 392003, Tomakomai-Shi
  - Investigational Site Number 392074, Urasoe-Shi
  - Investigational Site Number 392079, Urayasu-Shi
  - Investigational Site Number 392048, Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 40 centers in Japan. A total of 117 participants were screened between 23 February 2015 and 9 September 2015, 26 of whom were screen failures.
Pre-assignment Details: A total of 91 participants were randomized to receive monotherapy stratum (in a ratio of 1:1 to sarilumab 150 mg, once in every two weeks [q2w] or sarilumab 200 mg, q2w) or combination stratum (background non-methotrexate disease modifying anti-rheumatic drugs [Non-MTX DMARDs] along with sarilumab 150/ 200 mg q2w in 1:1 ratio).
Groups:
- Sarilumab 150 mg q2w + DMARDs: Participants received sarilumab 150 mg, subcutaneous (SC) injection, q2w along with non-MTX DMARDs for up to 52 weeks.
- Sarilumab 200 mg q2w + DMARDs: Participants received sarilumab 200 mg, SC injection, q2w along with non-MTX DMARDs for up to 52 weeks.
Period: Overall Study
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Started | 15 | 15 | 30 | 31
Completed | 13 | 9 | 27 | 30
Not Completed | 2 | 6 | 3 | 1
Not completed — Adverse Event | 2 | 5 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least one dose of investigational medicinal product (IMP), irrespective of compliance with the study protocol and procedures.
Groups:
- Sarilumab 150 mg q2w + DMARDs: Participants received sarilumab 150 mg, SC injection, q2w along with non-MTX DMARDs for up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w | Total
Number analyzed (Participants) | 15 | 15 | 30 | 31 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.9) | 63.3 (10.6) | 54.4 (13.8) | 52.5 (10.3) | 55.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 27 | 26 | 78
  Male | 3 | 2 | 3 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant who received IMP and did not necessary have to had a causal relationship with treatment. All AEs that occurred from the first dose of the IMP administration up to 6 weeks after last dose of treatment (up to Week 58) were considered as TEAEs. SAEs were AEs resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or a medically important event. TEAEs included both SAEs and non-SAEs.
Time Frame: Baseline up to Week 58
Population: Safety population included all randomized participants who actually received at least one dose or a partial dose of IMP analyzed according to the treatment actually received.
Measure: Number; unit: participants
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 15 | 15 | 30 | 31
participants
  Any TEAE | 14 | 13 | 25 | 28
  SAE | 0 | 3 | 1 | 2

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Abnormalities
Description: Criteria for potentially clinically significant vital sign abnormalities:
  * Systolic blood pressure (SBP) supine: <=95 mmHg and decrease from baseline (DFB) >=20 mmHg; >=160 mmHg and increase from baseline (IFB) >=20 mmHg
  * Diastolic blood pressure (DBP) supine: <=45 mmHg and DFB >=10 mmHg; >=110 mmHg and IFB ≥10 mmHg
  * SBP (Orthostatic): <=-20 mmHg
  * DBP (Orthostatic): <=-10 mmHg
  * Heart rate (HR) supine: <=50 beats per minute (bpm) and DFB >=20 bpm; >=120 bpm and IFB >=20 bpm
  * Weight: >=5% DFB; >=5% IFB
Time Frame: Baseline up to Week 58
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 15 | 15 | 30 | 31
participants
  SBP (supine) <=95 mmHg and DFB >=20 mmHg | 0 | 0 | 0 | 0
  SBP (supine) >=160 mmHg and IFB >=20 mmHg | 1 | 1 | 1 | 1
  DBP (supine) <=45 mmHg and DFB >=10 mmHg | 0 | 0 | 0 | 0
  DBP (supine) >=110 mmHg and IFB >=10 mmHg | 0 | 0 | 0 | 0
  SBP (orthostatic) <=-20 mmHg | 8 | 5 | 5 | 9
  DBP (orthostatic) <=-10 mmHg | 3 | 3 | 5 | 10
  HR (supine) <=50 bpm and DFB >= 20 bpm | 0 | 0 | 1 | 1
  HR (supine) >=120 bpm and IFB >=20 bpm | 0 | 0 | 0 | 0
  Weight >=5% DFB | 1 | 1 | 2 | 0
  Weight >=5% IFB | 3 | 2 | 12 | 7

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for potentially clinically significant ECG abnormalities:
  * PR Interval: >200 milliseconds (ms); >200 ms and IFB >=25%; >220 ms; >220 ms and IFB >=25%; >240 ms; >240 ms and IFB >=25%
  * QRS Interval: >110 ms; >110 ms and IFB >=25%; >120 ms; >120 ms and IFB >=25%
  * QT Interval: >500 ms
  * QTc Bazett (QTc B): >450 ms; >480 ms; >500 ms; IFB >30 and <=60 ms, IFB >60 ms
  * QTc Fridericia (QTc F): >450 ms; >480 ms; >500 ms; IFB >30 and <=60 ms; IFB >60 ms
Time Frame: Baseline up to Week 58
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 15 | 15 | 30 | 31
participants
  PR >200 ms | 0 | 0 | 0 | 1
  PR >200 ms and IFB >=25%: number analyzed (Participants) | 15 | 15 | 30 | 30
  PR >200 ms and IFB >=25% | 0 | 0 | 0 | 0
  PR >220 ms | 0 | 0 | 0 | 1
  PR >220 ms and IFB >=25%: number analyzed (Participants) | 15 | 15 | 30 | 30
  PR >220 ms and IFB >=25% | 0 | 0 | 0 | 0
  PR >240 ms | 0 | 0 | 0 | 0
  PR >240 ms and IFB >=25%: number analyzed (Participants) | 15 | 15 | 30 | 30
  PR >240 ms and IFB >=25% | 0 | 0 | 0 | 0
  QRS >110 ms | 0 | 2 | 0 | 1
  QRS >110 ms and IFB >=25%: number analyzed (Participants) | 15 | 15 | 30 | 30
  QRS >110 ms and IFB >=25% | 0 | 0 | 0 | 0
  QRS >120 ms | 0 | 2 | 0 | 0
  QRS >120 ms and IFB >=25%: number analyzed (Participants) | 15 | 15 | 30 | 30
  QRS >120 ms and IFB >=25% | 0 | 0 | 0 | 0
  QT >500 ms | 0 | 0 | 0 | 1
  QTc B >450 ms | 2 | 1 | 6 | 10
  QTc B >480 ms | 0 | 1 | 0 | 1
  QTc B >500 ms | 0 | 0 | 0 | 0
  QTc B IFB >30 and <=60 ms: number analyzed (Participants) | 15 | 15 | 30 | 30
  QTc B IFB >30 and <=60 ms | 0 | 1 | 2 | 1
  QTc B IFB >60 ms: number analyzed (Participants) | 15 | 15 | 30 | 30
  QTc B IFB >60 ms | 0 | 0 | 0 | 0
  QTc F >450 ms | 2 | 1 | 2 | 6
  QTc F >480 ms | 0 | 0 | 0 | 1
  QTc F >500 ms | 0 | 0 | 0 | 0
  QTc F IFB >30 and <=60 ms: number analyzed (Participants) | 15 | 15 | 30 | 30
  QTc F IFB >30 and <=60 ms | 0 | 0 | 0 | 0
  QTc F IFB >60 ms: number analyzed (Participants) | 15 | 15 | 30 | 30
  QTc F IFB >60 ms | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Hematological Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Hemoglobin: <=115 g/L (Male[M]) or <=95 g/L (Female[F]); >=185 g/L (M) or >=165 g/L (F); DFB >=20 g/L
  * Hematocrit: <=0.37 v/v (M) or <=0.32 v/v (F); >=0.55 v/v (M) or >=0.5 v/v (F)
  * Red blood cells (RBC): >=6 Tera/L
  * Platelets: <50 Giga/L; >=50 and <100 Giga/L; >=700 Giga/L
  * White blood cells (WBC): <3.0 Giga/L (Non-Black [NB]) or <2.0 Giga/L (Black [B]); >=16.0 Giga/L
  * Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B); <1.0 Giga/L
  * Lymphocytes: <0.5 Giga/L; >=0.5 Giga/L and <lower limit of normal (LLN); >4.0 Giga/L
  * Monocytes: >0.7 Giga/L
  * Basophils: >0.1 Giga/L
  * Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN >=0.5 Giga/L)
Time Frame: Baseline up to Week 58
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 15 | 15 | 30 | 31
participants
  Hemoglobin <=115 g/L (M) or <=95 g/L (F) | 0 | 1 | 1 | 3
  Hemoglobin >=185 g/L (M) or >=165 g/L (F) | 0 | 0 | 0 | 0
  Hemoglobin DFB >=20 g/L | 0 | 0 | 0 | 2
  Hematocrit <=0.37 v/v (M) or <=0.32 v/v (F) | 0 | 3 | 2 | 6
  Hematocrit >0.55 v/v (M) or >=0.5 v/v (F) | 0 | 0 | 0 | 0
  RBC >=6 Tera/L | 0 | 0 | 0 | 0
  Platelets <50 Giga/L | 0 | 0 | 0 | 0
  Platelets >=50 and <100 Giga/L | 1 | 1 | 1 | 0
  Platelets >=700 Giga/L | 0 | 0 | 0 | 0
  WBC <3.0 Giga/L (NB) or <2.0 Giga/L (B) | 6 | 9 | 7 | 9
  WBC >=16.0 Giga/L | 0 | 0 | 0 | 0
  Neutrophils <1.5 Giga/L (NB) or <1.0 Giga/L (B) | 8 | 11 | 8 | 13
  Neutrophils <1.0 Giga/L | 5 | 3 | 2 | 4
  Lymphocytes <0.5 Giga/L | 0 | 0 | 0 | 1
  Lymphocytes >=0.5 Giga/L and <LLN | 3 | 4 | 3 | 8
  Lymphocytes >4.0 Giga/L | 0 | 1 | 0 | 0
  Monocytes >0.7 Giga/L | 1 | 0 | 3 | 2
  Basophils >0.1 Giga/L | 1 | 0 | 0 | 5
  Eosinophils >0.5 Giga/L or >ULN (ULN >=0.5 Giga/L) | 0 | 0 | 2 | 2

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20, 50 and 70 Responses at Week 52
Description: ACR response is a composite rating scale that includes 7 variables: tender joints count (TJC [68 joints]); swollen joints count (SJC [66 joints]); levels of an acute phase reactant (high sensitivity C-reactive protein [hs-CRP level]); participant's assessment of pain (measured on 0 [no pain]-100 mm [worst pain] visual analog scale [VAS]); participant's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); physician's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); participant's assessment of physical function (measured by Health Assessment Question-Disability Index [HAQ-DI], with scoring range of 0 [better health] - 3 [worst health]). ACR20/50/70 response is defined as at least 20/50/70% improvement in both TJC and SJC, and at least 20/50/70% improvement in at least 3 of the 5 other assessments, respectively.
Time Frame: Week 52
Population: mITT population included all randomized participants who received at least one dose of IMP, irrespective of compliance with the study protocol and procedures.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 15 | 15 | 30 | 31
percentage of participants
  ACR20 | 73.3 | 40.0 | 76.7 | 74.2
  ACR50 | 60.0 | 33.3 | 56.7 | 54.8
  ACR70 | 53.3 | 26.7 | 26.7 | 25.8

6. Secondary Outcome: Change From Baseline at Week 52 in Disease Activity Score for 28 Joints Based on C-Reactive Protein (DAS28-CRP)
Description: DAS28-CRP is a composite score that contains 4 variables: TJC (based on 28 joints), SJC (based on 28 joints), participant's assessment of general health on VAS (range 0 [very well] to 100 mm [extremely bad]) and CRP (mg/L). DAS28-CRP total score ranges from 2-10 with a lower score indicating less disease activity. A DAS28-CRP above 5.1 indicates high disease activity, whereas below 3.2 indicates low disease activity and below 2.6 as disease remission.
Time Frame: Baseline, Week 52
Population: mITT population included all randomized participants who received at least one dose of IMP, irrespective of compliance with the study protocol and procedures. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 14 | 10 | 28 | 30
units on a scale | -2.90 (1.06) | -2.47 (0.84) | -2.62 (1.12) | -2.64 (1.35)

7. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 52
Description: HAQ-DI assessed the degree of difficulty participants experienced in 8 daily living activity domains during a week: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consisted of 2-3 items. Each items's difficulty was scored from 0-3 (0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do). Overall HAQ-DI score was computed as the sum of domain scores divided by the number of domains answered, providing a score from 0-3. Low scores denoted improvement of disability/lower degree of domain difficulty.
Time Frame: Baseline, Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 14 | 10 | 28 | 30
units on a scale | -0.52 (0.45) | -0.34 (0.60) | -0.48 (0.58) | -0.38 (0.34)

8. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Metabolic Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Glucose: <=3.9 mmol/L and <LLN; >=11.1 mmol/L (unfasted [unfas]) or >=7 mmol/L (fasted [fas])
  * Hemoglobin A1c (HbA1c): >8%
  * Total cholesterol: >=6.2 mmol/L; >=7.74 mmol/L
  * LDL cholesterol: >=4.1 mmol/L; >=4.9 mmol/L
  * Triglycerides: >=4.6 mmol/L; >=5.6 mmol/L
Time Frame: Baseline up to Week 58
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 15 | 15 | 30 | 31
participants
  Glucose <=3.9 mmol/L and <LLN | 0 | 0 | 1 | 1
  Glucose >=11.1 mmol/L (unfas) or >=7 mmol/L (fas) | 0 | 1 | 0 | 2
  HbA1c >8% | 0 | 0 | 0 | 1
  Total Cholesterol >=6.2 mmol/L | 6 | 7 | 12 | 13
  Total Cholesterol >=7.74 mmol/L | 1 | 1 | 1 | 2
  LDL Cholesterol >=4.1 mmol/L | 1 | 3 | 6 | 3
  LDL Cholesterol >=4.9 mmol/L | 0 | 1 | 2 | 1
  Triglycerides >=4.6 mmol/L | 0 | 0 | 0 | 1
  Triglycerides >=5.6 mmol/L | 0 | 0 | 0 | 1

9. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Electrolytes
Description: Criteria for potentially clinically significant abnormalities:
  * Sodium: <=129 mmol/L; >=160 mmol/L
  * Potassium: <3 mmol/L; >=5.5 mmol/L
  * Chloride: <80 mmol/L; >115 mmol/L
Time Frame: Baseline up to Week 58
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 15 | 15 | 30 | 31
participants
  Sodium <=129 mmol/L | 0 | 0 | 0 | 0
  Sodium >=160 mmol/L | 0 | 0 | 0 | 0
  Potassium <3 mmol/L | 0 | 0 | 0 | 0
  Potassium >=5.5 mmol/L | 0 | 0 | 0 | 0
  Chloride <80 mmol/L | 0 | 0 | 0 | 0
  Chloride >115 mmol/L | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Renal Function Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Creatinine: >=150 micromol/L (adults); >=30% change from baseline, >=100% change from baseline
  * Creatinine clearance: <15 mL/min; >=15 to <30 mL/min; >=30 to <60 mL/min; >=60 to <90 mL/min
  * Blood urea nitrogen: >=17 mmol/L
  * Uric acid: <120 micromol/L; >408 micromol/L
Time Frame: Baseline up to Week 58
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 15 | 15 | 30 | 31
participants
  Creatinine >=150 micromol/L (Adults) | 0 | 0 | 0 | 1
  Creatinine >=30% change from baseline | 3 | 3 | 6 | 5
  Creatinine >=100% change from baseline | 0 | 0 | 0 | 0
  Creatinine Clearance <15 mL/min | 0 | 0 | 0 | 0
  Creatinine clearance >=15 to <30 mL/min | 0 | 0 | 0 | 0
  Creatinine clearance >=30 to <60 mL/min | 6 | 6 | 6 | 5
  Creatinine clearance >=60 to <90 mL/min | 8 | 7 | 15 | 17
  Blood Urea Nitrogen >=17 mmol/L | 0 | 0 | 0 | 0
  Uric acid <120 micromol/L | 0 | 1 | 0 | 0
  Uric acid >408 micromol/L | 1 | 1 | 2 | 4

11. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Liver Function Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Alanine Aminotransferase (ALT): >1 ULN and <=1.5 ULN; >1.5 ULN and <=3 ULN; >3 ULN and <=5 ULN; >5 ULN and <=10 ULN; >10 ULN and <=20 ULN; >20 ULN
  * Aspartate aminotransferase (AST): >1 ULN and <=1.5 ULN; >1.5 ULN and <=3 ULN; >3 ULN and <=5 ULN; >5 ULN and <=10 ULN; >10 ULN and <=20 ULN; >20 ULN
  * Alkaline phosphatase: >1.5 ULN
  * Total bilirubin (TBILI): >1.5 ULN; >2 ULN
  * Conjugated bilirubin(CBILI): >1.5 ULN
  * Unconjugated bilirubin: >1.5 ULN
  * ALT >3 ULN and TBILI >2 ULN
  * CBILI >35% TBILI and TBILI >1.5 ULN
  * Albumin: <=25 g/L
Time Frame: Baseline up to Week 58
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 15 | 15 | 30 | 31
participants
  ALT >1 ULN and <=1.5 ULN | 3 | 4 | 7 | 6
  ALT >1.5 ULN and <=3 ULN | 2 | 1 | 3 | 2
  ALT >3 ULN and <=5 ULN | 1 | 0 | 1 | 4
  ALT >5 ULN and <=10 ULN | 1 | 0 | 0 | 0
  ALT >10 ULN and <=20 ULN | 0 | 0 | 0 | 0
  ALT >20 ULN | 0 | 0 | 0 | 0
  AST >1 ULN and <=1.5 ULN | 6 | 5 | 8 | 4
  AST >1.5 ULN and <=3 ULN | 1 | 0 | 2 | 3
  AST >3 ULN and <=5 ULN | 1 | 0 | 0 | 1
  AST >5 ULN and <=10 ULN | 0 | 0 | 0 | 0
  AST >10 ULN and <=20 ULN | 0 | 0 | 0 | 0
  AST >20 ULN | 0 | 0 | 0 | 0
  Alkaline Phosphatase >1.5 ULN | 0 | 0 | 0 | 0
  TBILI >1.5 ULN | 1 | 1 | 0 | 0
  TBILI >2 ULN | 0 | 0 | 0 | 0
  CBILI >1.5 ULN | 0 | 0 | 0 | 0
  Unconjugated Bilirubin >1.5 ULN | 0 | 0 | 0 | 0
  ALT> 3 ULN and TBILI >2ULN | 0 | 0 | 0 | 0
  CBILI >35% TBILI and TBILI >1.5 ULN | 0 | 0 | 0 | 0
  Albumin <=25 g/L | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form until the end of the study (Week 58) regardless of seriousness or relationship to IMP.
Description: Reported AEs are treatment-emergent AEs that developed/worsened during the 'on treatment period' (from the first IMP administration up to the 6 week after last IMP administration [up to Week 58]).
Groups:
- Sarilumab 150 mg q2w Monotherapy: Participants received sarilumab 150 mg, SC injection, q2w for up to 52 weeks.
- Sarilumab 200 mg q2w Monotherapy: Participants received sarilumab 200 mg, SC injection, q2w for up to 52 weeks.
Arm/Group | Sarilumab 150 mg q2w + DMARDs | Sarilumab 200 mg q2w + DMARDs | Sarilumab 150 mg q2w Monotherapy | Sarilumab 200 mg q2w Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/15 | 3/15 | 1/30 | 2/31
Other Adverse Events (participants affected / at risk) | 14/15 | 13/15 | 22/30 | 23/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab 150 mg q2w + DMARDs (N=15) | Sarilumab 200 mg q2w + DMARDs (N=15) | Sarilumab 150 mg q2w Monotherapy (N=30) | Sarilumab 200 mg q2w Monotherapy (N=31)
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 0 | 1 | 0
Periorbital abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab 150 mg q2w + DMARDs (N=15) | Sarilumab 200 mg q2w + DMARDs (N=15) | Sarilumab 150 mg q2w Monotherapy (N=30) | Sarilumab 200 mg q2w Monotherapy (N=31)
Neutropenia (Blood and lymphatic system disorders) | 5 | 3 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 4 | 3 | 4
Injection site erythema (General disorders) | 0 | 1 | 1 | 6
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 | 1 | 1
Injection site rash (General disorders) | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 2
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1 | 4
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 5 | 13 | 14
Periodontitis (Infections and infestations) | 0 | 1 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 2 | 1
Protein urine (Investigations) | 0 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.